CLINICAL TRIAL: NCT03075735
Title: Prospective Multicentre Cohort Study of the Prevalence and Clinical Impact of Germline Deleterious Mutations in DNA Repair Genes of Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Prospective Multicentre Cohort Study PROREPAIR-B (mCRPC)
Status: Completed | Type: Observational
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other); Instituto de Investigacion Biomedica de Malaga (Other)
Responsible Party: Sponsor
Other Study IDs: CNIO-CP-2013-02-B
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Castration-Resistant Prostate Cancer; DNA-repair; BRCA1; BRCA2; ATM; PALB2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, archival FFPE and fresh tumour samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic castration resistant patients: The exposition to the primary analysis risk factor (germline deleterious mutation in BRCA1, BRCA2, ATM or PALB2 gene) will be determined after inclusion. Briefly, a NGS targeted-panel based on the majority of genes included in the BROCA panel and additional DNA-repair related genes has been designed based on the available technology. The pathogenicity of germline variants will be determined according to established American College of Medical Genetics and Genomics and Association for Molecular Pathology current consensus at the time of final primary outcome analyses. Variants will also be reviewed against published literature and public databases. According to their mutation-carrier status patients will be classified as: A) Mutation Carriers in BRCA1, BRCA2, ATM and PALB2 genes; B) Mutation carriers in other genes included in the BROCA panel; C) Mutation carriers in others DNA-repair genes D)Non-carriers

SUMMARY:
PROREPAIR is a prospective multicenter observational cohort study of unselected patients with metastatic Castration Resistant Prostate Cancer (mCRPC) with unknown germline mutational status at study entry and who are candidates to start 1st line treatment with any approved survival-prolonging agent.

The study aims to evaluate the impact of aberrations in DNA-repair genes,(BRCA1, BRCA2, ATM and PALB2 and other genes) on cause-specific survival from the diagnosis of the metastatic castration resistant status and other outcomes.

DETAILED DESCRIPTION:
This is a non-interventional study in which eligible patients are prospectively followed-up until death or the end-of-study, whichever happens first.

Patients are enrolled after mCRPC diagnosis and before or within the 6 first months of starting a first-line treatment with any approved survival-prolonging agent for mCRPC. First and subsequent treatment lines will be chosen according to the patients and their treating physicians preferences and will not be dictated by this study.

A whole blood sample for germline DNA extraction as well as any available archival prostate cancer tissue samples will be collected at baseline. Optional plasma, serum and whole blood samples will be collected at baseline and at different time points along the evolution of the disease. A sample will be collected within the last 6 months of life.

Survival and treatment outcomes including biochemical, radiological and clinical progression with standard approved agents abiraterone, enzalutamide, docetaxel, cabazitaxel and radium-223 will be prospectively collected.

Primary aim is to evaluate the prevalence and impact of DNA repair germline mutations in the BRCA1, BRCA2, ATM and PALB2 genes on cause-specific survival from mCRPC. Secondary aims will include the correlation of additional germline alterations in DNA-repair with survival and treatment outcomes; the analyses of the survival and treatment outcomes impact of somatic alterations in these genes and the role of germline and somatic defects in the clonal evolution of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent.
2. Patients must be ≥18 years old.
3. Histologically confirmed prostate cancer
4. presence of metastatic disease according to Bone-, CT- and/or MRI-scan.
5. Confirmed castration resistant prostate cancer defined as disease progression despite castrate levels of testosterone (<0.5ng/mL) and either a continuous rise in the serum prostate-specific antigen (PSA) levels, the progression of preexisting disease and /or the appearance of new metastases. Patients must be maintained on aLHRH or have underwent bilateral orchiectomy.
6. Eligible patients are due to start or have started first-line treatment with any approved survival-prolonging therapy for mCRPC within a period of 6 months from study entry.
7. ECOG performance status ≤21.
8. Unknown mutation carrier status at the study entry.

Exclusion Criteria:

1. Previous cancer diagnosis, except those patients who had a localized malignant tumour and who are five years cancer-free or those diagnosed with skin cancers (of non-melanoma type) or excised in situ carcinomas.
2. Any prior medical history that according to the judgement of the investigator might interfere with the subject´s granting of informed consent or the safe execution of the procedures required in the study.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed castration resistant prostate cancer without known mutation carrier status at study entry
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the impact of BRCA1, BRCA2, ATM, PALB2 germline mutations | 42 months
  To assess the impact of BRCA1, BRCA2, ATM, PALB2 germline mutations on cause-specific survival from diagnosis of metastatic castration resistance status.

SECONDARY OUTCOMES:
Analysis of the impact of other germline mutations in other DNA repair genes | 42 months
  To analyze the impact of other germline mutations in other DNA repair genes on cause-specific survival from diagnosis of metastatic castration resistance
Correlation between DNA repair germline mutation carrier status and survival | 42 months
  To explore the correlation between DNA repair germline mutation carrier status and cause-specific survival following first, second, third and successive treatment lines.
Correlation between DNA repair germline mutation and biochemical response | 42 months
  To study the correlation between BRCA1, BRCA2, ATM, PALB2 and other genes mutation carrier status and the biochemical response and time to biochemical progression following treatment with abiraterone acetate, enzalutamide, radium-223, docetaxel and/or cabazitaxel.
Correlation between DNA repair germline mutation and radiographic response | 42 months
  To study the correlation between BRCA1, BRCA2, ATM, PALB2 and other genes mutation carrier status and the radiographic response and time to radiographic progression following treatment with abiraterone acetate, enzalutamide, radium-223, docetaxel and/or cabazitaxel.
Correlation between somatic DNA repair abnormalities with cause-specific survival | 42 months
  To explore in this cohort the correlation between somatic DNA repair abnormalities with cause-specific survival and other treatment-related outcomes.
Correlation between DNA repair somatic and germline alterations with prior prostate cancer history | 42 months
  To correlate DNA repair somatic and germline alterations with prior prostate cancer history characteristics and established risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: David Olmos, MD, Principal Investigator — Centro Nacional de Investigaciones Oncologicas CARLOS III

IPD SHARING:
Plan to Share IPD: No